CLINICAL TRIAL: NCT05649709
Title: Fourteen-day Vonoprazan and Low-or High-dose Amoxicillin Dual Therapy for Eradicating Helicobacter Pylori Infection: a Prospective, Multi-centers, Open-labeled, Non-inferior, Randomized Clinical Study
Brief Title: Helicobacter Pylori and Vonoprazan Dual Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Iv Nonghua, Professor, The First Affiliated Hospital of Nanchang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hp therapy of NCU
Record Dates: First submitted 2022-11-27; First posted 2022-12-14 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Helicobacter Pylori
Keywords: Helicobacter pylori; vonoprazan; amoxicillin; eradication

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- vonoprazan and low-dose amoxicillin dual therapy (Experimental): 1000 mg amoxicillin capsules twice daily and 20 mg vonoprazan Fumarate Tablets twice daily for 14 days
  Interventions: Drug: L-VA dual therapy
- vonoprazan and high-dose amoxicillin dual therapy (Active Comparator): 1000mg amoxicillin capsules three times daily and 20mg vonoprazan Fumarate Tablets twice daily for 14 days
  Interventions: Drug: H-VA dual therapy

INTERVENTIONS:
Drug: L-VA dual therapy — 1000mg amoxicillin capsules twice times daily and 20mg vonoprazan Fumarate Tablets twice daily for 14 days
  Other Names: L-VA
  Arms: vonoprazan and low-dose amoxicillin dual therapy
Drug: H-VA dual therapy — 1000mg amoxicillin capsules three times daily and 20mg vonoprazan Fumarate Tablets twice daily for 14 days
  Other Names: H-VA
  Arms: vonoprazan and high-dose amoxicillin dual therapy

SUMMARY:
Our previous study included 119 Helicobacter pylori(H. pylori)-infected Chinese patients without previous eradication history who were randomized to low-or high-dose amoxicillin-vonoprazan regimens consisting of amoxicillin 1 gram either b.i.d. or t.i.d plus vonoprazan 20 mg b.i.d for 7 or 10 days. Neither 7-or 10-day VA dual therapy with either b.i.d. or t.i.d. amoxicillin achieved satisfied efficacy (i.e., <90%) when given as first-line treatment for H. pylori infection. This study evaluated the efficacy and safety of low-and high-dose amoxicillin-vonoprazan dual therapy for 14 days as first-line treatment for H. pylori in China.

DETAILED DESCRIPTION:
Upper gastrointestinal endoscopy examinations were performed for all participants and biopsies from gastric antrum and body were obtained. All the collected gastric biopsy specimens were sent to Jiangxi Provincial Key Laboratory of Digestive Diseases, First Affiliated Hospital of Nanchang University for susceptibility testing of antibiotics. The minimum inhibitory concentrations of antibiotics (amoxicillin, metronidazole, clarithromycin, levofloxacin and tetracycline) were determined by E-test. The inhibition zone for furazolidone was determined by the Kirby-Bauer disc diffusion method. Detailed procedure for detecting antibiotics resistance were consistent with our previous study. A strain was considered as resistant if minimum inhibitory concentration >0.125 μg/mL for amoxicillin, >8 μg/mL for metronidazole, ≥1 μg/mL for clarithromycin, >2 μg/mL for levofloxacin, ≥2 μg/mL for tetracycline, the inhibition zone was ≤7mm for furazolidone.

The detailed demographics and characteristics (sex, age, nationality, height, weight, education status, dwelling area, history of smoking and alcohol etc.) were recorded. The treatment-related adverse events (TEAEs) were recorded. We defined adherence as good if the participants took ≥80% drugs of the regimen during the consecutive 14 days. The H. pylori status after therapy was evaluated by ¹³C-UBT at least 6 weeks after completion of treatment. Proton pump inhibitors and antibiotics were stopped at least 2 and 4 weeks before ¹³C-UBT, respectively.

The stool samples were collected at baseline (before treatment), week 2 (after eradication) and week 8-10 (confirmation of H. pylori status). We sent the stool samples from subjects with successful eradication for metagenome DNA extraction and shotgun sequencing to avoid the influence of H. pylori eradication failure on gut microbiota. Briefly, OMEGA Mag-Bind Soil DNA Kit (Omega Bio-Tek, Norcross, GA, USA) was used to extract total microbial genomic DNA samples. Metagenome shotgun sequencing libraries from extracted microbial DNA was constructed by Illumina TruSeq Nano DNA LT Library Preparation Kit, which was then sequenced by Illumina NovaSeq platform (Illumina, USA) with PE150 strategy at Personal Biotechnology Co., Ltd. (Shanghai, China).

Raw sequencing reads were subjected to processing to yield quality-filtered reads suitable for further analysis, including removal of adapter and low-quality reads. Subsequently, minimap2 was utilized to align reads to the host genome of human and eliminate host contamination. Gene prediction was carried out on the generated contigs from each sample, whose translated protein sequences were subsequently pooled and clustered using mmseqs2. The lowest common ancestor taxonomy of the non-redundant genes was ascertained using mmseqs2 in "taxonomy" mode, by aligning them against a customized database comprising protein sequences of bacteria from GTDB (release 207: https://data.ace.uq.edu.au/public/gtdb/data/releases/), fungi from NCBI-nr (https://ftp.ncbi.nlm.nih.gov/blast/db/FASTA/), and viruses from RVDB (version 24.1: https://rvdb.dbi.udel.edu/download/). In order to assess the abundance of genes, high-quality reads from each sample were mapped onto the contigs using minimap2 and read counts were computed using htseq. Abundance values in metagenomes were normalized using copies per kilobase per million mapped reads. Clean high-quality reads were processed and profiled with ARGs-OAP (version 2.0) by querying against the SARG (version 3.0-F) database, which is a structural antimicrobial resistance genes database containing 32 types and 2842 subtypes of antibiotic resistance genes. In order to perform the quantification and downstream analysis of diversity indices, resistome profiling, and prevalence ranking, the abundance of antibiotic resistance genes at type and subtype level were normalised to the number of 16S rRNA genes.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive H. pylori-infected subjects ages from 18 to 70 without eradication history

Exclusion Criteria:

* allergy to amoxicillin or vonoprazan;
* acute upper gastrointestinal bleeding, gastric cancer or other tumors, Zollinger-Ellison syndrome, history of gastric surgery;
* serious illness including neurological, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urological, endocrinological or hematological disorders;
* pregnancy or breast feeding;
* proton pump inhibitors and antibiotics use within one month;
* not willing to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
The efficacy of VA dual therapy | 6-8 weeks after treatment
  The confirmation of H. pylori status was evaluated by urea breath test

SECONDARY OUTCOMES:
treatment-emergent adverse events | 1 day after eradication
  the frequency and severity of treatment-emergent adverse events
compliance | 1 day after eradication
  good compliance was defined as achieving ≥80% of drugs included in the regimes and bad compliance was defined as achieving <80% drugs.
resistance of antibiotics | before the eradication
  An E-test was used to determine the minimum inhibitory concentrations (MIC) of Amoxicillin (AMO), Metronidazole (MET), Clarithromycin (CLA), Levofloxacin (LEV) and tetracycline (TET). The Kirby-Bauer disc diffusion method (Oxoid) was used to determine the inhibition zone for Furazolidone (FUR). A strain was considered resistant if the MIC>1 mg/mL for AMO, ≥1 mg/mL for CLA, >2 mg/mL for TET, >4 mg/mL for MET, MIC >1 mg/mL for LEV and if the inhibition zone was <7 mm for FUR. H. pylori strain ATCC 43504 was included as an antibiotic susceptibility testing qualitycontrol. All antibiotic susceptibility tests were conducted at the Institute of Gastroenterology and Hepatology, First Affiliated Hospital of Nanchang University.
the alteration of gut microbiota | before eradication，1 day after eradication and confirmation（6-8 weeks after treatment）
  The fecal samples were collected before eradication,1 day after eradication and confirmation（6-8 weeks after treatment）. Bioinformatics of gut microbiome were performed using QIIME2 with slight modification and R packages. Briefly, Non-singleton ASVs were aligned and used to construct a phylogeny with fasttree2. Alpha-diversity metrics were calculated using the ASV table in QIIME2 and visualized as box plots. ASV-level ranked abundance curves were generated to compare the richness and evenness of ASVs among samples. Beta diversity analysis was conducted to explore the structural variation of microbial communities across samples using Bray-Curtis metrics and visualized via principal coordinate analysis (PCoA). The significance of microbiota structure differences among groups was assessed by Permanova using QIIME2. Microbial functions were predicted by PICRUSt2 upon KEGG (https://www.kegg.jp/) databases.

CONTACTS AND LOCATIONS:
Overall Officials: Nong-Hua Lu, phD, Principal Investigator — The First Affiliated Hospital of Nanchang University
Locations (1):
- The First Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu Y, Zhang ZY, Wang F, Zhuang K, Xu X, Liu DS, Fan HZ, Yang L, Jiang K, Zhang DK, Xu L, Tang JH, Liu XM, He C, Shu X, Xie Y, Lau JYW, Zhu Y, Du YQ, Graham DY, Lu NH. Effects of amoxicillin dosage on cure rate, gut microbiota, and antibiotic resistome in vonoprazan and amoxicillin dual therapy for Helicobacter pylori: a multicentre, open-label, non-inferiority randomised controlled trial. Lancet Microbe. 2025 Mar;6(3):100975. doi: 10.1016/j.lanmic.2024.100975. Epub 2024 Dec 18. PMID 39708826